CLINICAL TRIAL: NCT03092401
Title: Hepatopulmonary Syndrome and Postoperative Complications After Liver Transplantation : A Case-control Study.
Acronym: HPS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0210
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hepatopulmonary Syndrome; Liver Cirrhosis
Keywords: Liver transplantation; Hepatopulmonary Syndrome; Liver Cirrhosis
MeSH Terms: conditions — Hepatopulmonary Syndrome; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hepatic transplant patients with hepatopulmonary syndrome
- hepatic transplant patients without hepatopulmonary syndrome

SUMMARY:
Hepatopulmonary Syndrome is a respiratory complication of liver cirrhosis defined as a triad: hypoxemia (PaO2 < 80 mmHg in room air), chronic liver disease and intrapulmonary vasodilatations. Its prevalence varies between 4 and 32%. Numerous treatments have been tried but the only efficient therapy to cure the syndrome is liver transplantation. Without transplantation it is associated with a higher mortality which is the reason why hepatopulmonary syndrome patients have a higher priority to transplantation. However it appears in some restricted studies that hepatopulmonary syndrome is associated with more postoperative complications (infections, vascular and biliary complications, prolonged length of mechanical ventilation…).

The investigators hypothesised that hepatopulmonary syndrome patients have more postoperative complications after liver transplantation than non hepatopulmonary syndrome patients matched on age, MELD (Model for End-Stage Liver Disease) score, comorbidities, perioperative transfusion and noradrenaline doses.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplanted patients

Exclusion Criteria:

* Living donor transplantation
* Bipartition transplantation
* Non-heat-beating donor transplantation
* Minor
* Double or multiple organ transplantation
* Non cirrhotic patients
* Retransplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent liver transplantation between 2010 and 2016
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-03-31 (Estimated); Study Completion 2017-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rates in hepatic transplant patients with or without hepatopulmonary syndrome | 1 year post liver transplantation
  Collection of medical (cardiac, pulmonary, renal, infectious, neurological) and Surgical (vascular, digestive) complications in hepatic transplant patients with or without hepatopulmonary syndrome

SECONDARY OUTCOMES:
Length of Mechanical Ventilation | 1 year post liver transplantation
Length of ICU stay | 1 year post liver transplantation
Length of Hospital Stay | 1 year post liver transplantation
Delay of hepatopulmonary syndrome resolution | 1 year post liver transplantation